CLINICAL TRIAL: NCT03775291
Title: Fitbit Sleep Apnea Alert Software Validation Study
Brief Title: Validation of Software for Assessment of Sleep Apnea From Data Acquired by a Wearable Smartwatch
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fitbit LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 129-0318-01
Record Dates: First submitted 2018-12-03; First posted 2018-12-13 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low pre-test likelihood for sleep apnea: Subjects at low risk for having sleep apnea due to lack of known risk factors and no complaints of symptoms related to sleep apnea (e.g., excessive daytime sleepiness)
  Interventions: Diagnostic Test: Simultaneous assessment of sleep apnea by polysomnogram and wearable device
- High pre-test likelihood for sleep apnea: Suspected sleep apnea patients who are undergoing sleep tests as part of normal medical care or are also known to be non-compliant with therapy.
  Interventions: Diagnostic Test: Simultaneous assessment of sleep apnea by polysomnogram and wearable device

INTERVENTIONS:
Diagnostic Test: Simultaneous assessment of sleep apnea by polysomnogram and wearable device — Characterization of sleep apnea by lab-based polysomnogram

SUMMARY:
This clinical validation study aims to evaluate the utility of Fitbit's Sleep Apnea Alert software for minimally invasive monitoring of sleep apnea events to alert users of their risk of sleep apnea. The Sleep Apnea Alert software analyses data from a Fitbit commercially available wrist photoplethysmogram (PPG) device. The Sleep Apnea Alert software is an investigational software as medical device (SaMD) and is designed to retrospectively process data and flag users who have physiological signals consistent with an apnea-hypopnea index (AHI) of 15 or greater. This clinical validation study will be used to validate Fitbit's PPG-based sleep apnea algorithm. The outputs of the Fitbit Sleep Apnea Alert software will not be available to study participants, as the scope of this study is to gather validation data only and does not include testing product usability components.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent
* Comfortable reading the provided written study instructions in English (and/or local language) and using a smartphone in English (and/or local language).
* Have medical insurance either in the form of private insurance or a national health program.

Exclusion Criteria:

* No implanted cardiac devices
* Not pregnant. Pregnancy status will be confirmed per patient report of medical history, i.e., patients will be asked if they are pregnant or may be pregnant, and date of last menstrual cycle.
* No medical conditions which might lead to consistently low levels of perfusion in the vasculature at the wrist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects referred to sleep labs for a clinical evaluation or subjects with previous sleep apnea who are known to be non-compliant with treatment.
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of PSG-assessed AHI with multi-night estimate derived from wearable device. | Nightly basis averaged over 7 nights.
  Percent agreement between subjects classified as Apnea Hypopnea Index (AHI)≥15 or <15 as determined by a single night of lab based polysomnogram , versus the corresponding estimate (averaged over 7 nights) from the wearable device. [This primary outcome data will also be expressed as per-subject sensitivity and specificity of the wearable device to correctly identify subjects with AHI≥15 and AHI<15 respectively]

SECONDARY OUTCOMES:
Single night comparison between PSG and wearable device data on a per-subject basis | 1 night
  Percent agreement between subjects classified as Apnea Hypopnea Index (AHI)≥15 or <15 as determined by a single night of lab based polysomnogram , versus the corresponding estimate on the same night as PSG from the wearable device. [This primary outcome data will also be expressed as per-subject sensitivity and specificity of the wearable device to correctly identify subjects with AHI≥15 and AHI<15 respectively]
Single night comparison between PSG and wearable device data on a per-epoch basis | 1 night
  Percent agreement on a per one-minute epoch basis for the presence of sleep apnea between the polysomnogram and the corresponding simultaneous estimate from the wearable device .

CONTACTS AND LOCATIONS:
Overall Officials: Conor Heneghan, PhD, Study Director — Fitbit LLC
Locations (6):
- United States (5):
  - Jasper Summit Research, Jasper, Alabama
  - Peninsula Sleep Center, Burlingame, California
  - Sleep Center Orange County, Irvine, California
  - Neurotrials Inc, Atlanta, Georgia
  - SleepMed Inc, Columbia, South Carolina
- St Vincent's University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
No: There is not a plan to make IPD available.